CLINICAL TRIAL: NCT00331578
Title: Multi-Center Registry Trial of EXCEL Biodegradable Polymer Drug-Eluting Stent
Acronym: CREATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Medical Systems Ltd (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-06-6
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2009-01

CONDITIONS: AMI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Excel drug-eluting coronary artery stent

SUMMARY:
The trial aims to evaluate 12-month long-term efficiency of Excel stent in the treatment of coronary heart disease and inhibition of restenosis after coronary artery stenting as well as a 12 months' long-term safety after the cessation of clopidogrel as an anti-platelet drugs used for 6 months after the implantation of degradable drug coating stent.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who should be full fill the criteria of using Excel stent.
2. Each included patient should allowed to use Excel stent.
3. Complete revascularization can be achieved through one invasive operation.

Exclusion Criteria:

1. Patient do not suitable to use Excel stent, for example, not tolerant to anti-platelet drug or undergo cardiac/non-cardiac surgery recently.
2. Patient with multiple branch lesions, thus the single Excel stent cannot resolve the condition.
3. NYH Cardiac functional grading>3 or Echocardiography LVEF<0.3.
4. Patient with complete revascularization cannot be resolved by one operation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2077 (Actual)
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
MACE(Major adverse cardiac events) | 12 months

SECONDARY OUTCOMES:
MACE | 30 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Ph.D., Principal Investigator — Shenyang Northern Hospital

REFERENCES:
- [Derived] Li Y, Han Y, Zhang L, Jing Q, Wang X, Yan G, Ma Y, Wang G, Wang S, Chen X, Yang L, Zhu G, Liu H, Jiang T. Clinical efficacy and safety of biodegradable polymer-based sirolimus-eluting stents in patients with diabetes mellitus insight from the 4-year results of the create study. Catheter Cardiovasc Interv. 2013 Jun 1;81(7):1127-33. doi: 10.1002/ccd.24649. Epub 2013 Feb 26. PMID 22945767
- [Derived] Han Y, Jing Q, Xu B, Yang L, Liu H, Shang X, Jiang T, Li Z, Zhang H, Li H, Qiu J, Liu Y, Li Y, Chen X, Gao R; CREATE (Multi-Center Registry of Excel Biodegradable Polymer Drug-Eluting Stents) Investigators. Safety and efficacy of biodegradable polymer-coated sirolimus-eluting stents in "real-world" practice: 18-month clinical and 9-month angiographic outcomes. JACC Cardiovasc Interv. 2009 Apr;2(4):303-9. doi: 10.1016/j.jcin.2008.12.013. PMID 19463441